CLINICAL TRIAL: NCT07280455
Title: The Effectiveness of Gold Fixed Retainers Compared to Conventional Stainless Steel Retainers: A Randomized Clinical Trial
Brief Title: Effectiveness of Gold Fixed Retainers Compared to Conventional Stainless Steel Retainers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noor Sattar Raheem (Other)
Responsible Party: Sponsor-Investigator, Noor Sattar Raheem, Postgraduate Researcher (Principal Investigator), University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UOB-RCT-ORTHO-GOLDSS-2025
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Orthodontic Retention Appliance; Orthodontic Relapse
Keywords: fixed retainer; gold-coated retainer wire; stainless steel retainer wire; Little's Irregularity Index; retainer failure; periodontal indices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking is used for participants, outcome assessors, and the data analyst. The treating orthodontist (care provider) who places the fixed retainer cannot be blinded due to visible differences between the retainer wire types. Participants are not informed of group assignment. Outcome assessments are performed on coded study records/models by a blinded examiner, and the dataset is coded prior to statistical analysis, which is conducted by a blinded data analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gold-coated fixed retainer wire (Experimental): Participants will receive a mandibular canine-to-canine fixed retainer fabricated and bonded using the standardized protocol. The allocated device is a 0.0195-inch gold-plated multistranded wire (penta twist, five-strand).
  Interventions: Device: Gold-coated fixed retainer wire
- Stainless steel fixed retainer wire (Active Comparator): Participants will receive a mandibular canine-to-canine fixed retainer fabricated and bonded using the standardized protocol. The allocated device is a 0.0195-inch dead-soft multistranded stainless-steel wire (coaxial, six-strand).
  Interventions: Device: Stainless steel fixed retainer wire

INTERVENTIONS:
Device: Gold-coated fixed retainer wire — Participants will receive a bonded mandibular fixed retainer extending canine-to-canine. The retainer will be fabricated using a gold-coated retainer wire and bonded to the lingual surfaces of the mandibular anterior teeth using standard orthodontic bonding procedures. After placement, participants will be followed at scheduled visits (baseline and follow-ups at 1 month, 3 months, and 6 months) to evaluate clinical stability and retainer performance. At each follow-up visit, the retainer will be clinically examined for integrity, and any failure/complication events will be recorded (e.g., debonding/loosening, fracture, or need for repair). Clinical outcome assessments will include mandibular anterior alignment/stability (Little's Irregularity Index), periodontal indices, and occlusal assessment, Microbiological sampling will consist of plaque/swab samples collected at each follow-up visit.
  Arms: Gold-coated fixed retainer wire
Device: Stainless steel fixed retainer wire — Participants will receive a bonded mandibular fixed retainer extending canine-to-canine. The retainer will be fabricated using a conventional stainless steel retainer wire and bonded to the lingual surfaces of the mandibular anterior teeth using standard orthodontic bonding procedures. After placement, participants will be followed at scheduled visits (baseline and follow-ups at, 1 month, 3 months, and 6 months) to evaluate clinical stability and retainer performance. At each follow-up visit, the retainer will be clinically examined for integrity, and any failure/complication events will be recorded (e.g., debonding/loosening, fracture, or need for repair). Clinical outcome assessments will include mandibular anterior alignment/stability (Little's Irregularity Index), periodontal indices, and occlusal assessment. Microbiological sampling will consist of plaque/swab samples collected at each follow-up visit.
  Arms: Stainless steel fixed retainer wire

SUMMARY:
This randomized clinical trial will compare the effectiveness of a gold-plated multistranded mandibular fixed retainer versus a conventional multistranded stainless-steel fixed retainer in maintaining lower anterior tooth alignment after completion of orthodontic treatment. Eligible participants (post-orthodontic patients requiring mandibular fixed retention) will be allocated in a 1:1 ratio to receive either a gold-plated 0.0195-inch multistranded retainer or an identical-gauge 0.0195-inch stainless-steel multistranded retainer. Participants will be followed for 6 months.

The primary outcome is post-treatment stability of mandibular anterior alignment, assessed by changes in Little's Irregularity Index over time, along with retainer failure outcomes (e.g., time to first failure and tooth-level failure events). Secondary outcomes include periodontal health indices and related clinical measures collected at baseline and follow-up visits.

For the microbiological assessment, plaque/biofilm will be collected from the retainer using sterile swabs at 1 month, 3 months, and 6 months to evaluate bacterial levels associated with each retainer material.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15-30 years.
* Patients who have completed comprehensive orthodontic treatment ,with well-aligned mandibular anterior teeth (Little's Irregularity Index ≤ 0.5 mm) at debond; both extraction and non-extraction cases are eligible.
* Patients with good oral hygiene and healthy periodontium at baseline; no previous bonded retainer.
* All mandibular anterior teeth present (canine-canine), with sound lingual enamel suitable for bonding.

Exclusion Criteria:

* Patients with a history of rapid maxillary expansion (RME) or surgically assisted RME (SARME).
* Patients with a cleft lip / and or palate (craniofacial anomalies).
* Patients with marked deep overbite and/or parafunctional habits (e.g., bruxism, clenching).
* Patients with conditions precluding reliable bonding in the mandibular anterior segment (active caries, extensive restorations, enamel fractures) or missing teeth from canine to canine.
* Patients with medical/periodontal conditions likely to affect gingival health (e.g., active periodontitis, uncontrolled systemic disease).

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in mandibular incisor alignment (Little's Irregularity Index, ΔLII) | Baseline (T0) to 6 months after retainer placement (assessed at 1, 3, and 6 months)
  Little's Irregularity Index (LII) is a quantitative scale of mandibular anterior alignment, calculated as the sum of the linear displacements (in mm) of the contact points of the six mandibular anterior teeth. Scores range from 0 mm (perfect alignment, no irregularity) to ≥10 mm (very severe irregularity); higher scores indicate greater crowding and therefore a worse outcome.
  LII will be measured for the mandibular anterior teeth (canine-to-canine) at baseline (T0, before fixed-retainer placement) and at follow-up visits (T1 = 1 month, T2 = 3 months, T3 = 6 months). The primary endpoint is the change in LII (follow-up LII minus baseline LII), comparing gold-plated versus stainless-steel fixed-retainer groups.
Time to first fixed-retainer failure (survival) | From retainer placement to 6 months after placement.
  Time (days) from fixed retainer bonding to the first failure event requiring repair/rebonding/replacement. Failures will be recorded and classified (e.g., adhesive-enamel debond, wire-composite debond, wire fracture, partial/complete loosening) and compared between groups.

SECONDARY OUTCOMES:
Plaque accumulation at mandibular anterior teeth (Silness-Löe Plaque Index) | Baseline and 1, 3, and 6 months.
  Silness-Löe Plaque Index is a 4-point scale (0-3) that scores plaque accumulation on tooth surfaces adjacent to the gingival margin. Scores range from 0 (no plaque) to 3 (abundant soft deposits); higher scores indicate poorer oral hygiene and a worse periodontal condition. The mean Plaque Index will be recorded for the mandibular anterior teeth adjacent to the fixed retainer at baseline (T0, before retainer placement) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement, and compared between the gold-plated and stainless-steel fixed-retainer groups.
Microbiological plaque outcome | Follow-up visits at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement.
  Biofilm will be collected using a sterile swab moved along interdental spaces over the exposed retainer, then placed in transport medium and sent for cultivation. After incubation on agar, the total number of bacterial colonies (colony-forming units, CFU) will be counted for each sample. Higher CFU counts indicate greater plaque accumulation and a worse periodontal outcome. Samples will be collected at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement and compared between the gold-plated and stainless-steel fixed-retainer groups.
Change in mandibular inter-canine width | Baseline (T0, before retainer placement) and follow-up visits at 1 month (T1), 3 months (T2), and 6 months (T3).
  Mandibular inter-canine width (mm) will be measured on study casts/impressions as the linear distance between the cusp tips of the right and left mandibular canines. Measurements will be taken at baseline (T0, before fixed-retainer placement) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement. The outcome is the change in inter-canine width from baseline at each follow-up visit; larger absolute changes indicate greater relapse and worse post-treatment occlusal stability. Changes will be compared between the gold-plated and stainless-steel fixed-retainer groups.
Gingival inflammation at mandibular anterior teeth (Löe-Silness Gingival Index) | Baseline and 1, 3, and 6 months after retainer placement.
  Gingival condition will be assessed using the Löe-Silness Gingival Index, a 4-point scale (0-3) where 0 = normal gingiva, 1 = mild inflammation, 2 = moderate inflammation, and 3 = severe inflammation with ulceration and/or spontaneous bleeding. Higher scores indicate more severe gingival inflammation and a worse periodontal outcome. The mean Gingival Index will be recorded for the mandibular anterior teeth adjacent to the fixed retainer at baseline (T0) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement, and compared between the two retainer groups.
Probing pocket depth at mandibular anterior teeth | Baseline and 1, 3, and 6 months after retainer placement.
  Probing pocket depth (PPD) in millimeters will be measured at specified sites around the mandibular anterior teeth using a calibrated periodontal probe. Higher values indicate deeper pockets and a worse periodontal outcome. Mean PPD will be calculated for the mandibular anterior region at baseline (T0) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement, and compared between the two fixed-retainer groups.
Change in mandibular arch length | Baseline (T0, before retainer placement) and 1, 3, and 6 months (T1, T2, T3) after retainer placement.
  Mandibular arch length (mm) will be measured on study casts as the linear distance from the mesial surface of the right mandibular first permanent molar to the mesial surface of the left mandibular first permanent molar, parallel to the occlusal plane. Measurements will be taken at baseline (T0, before fixed-retainer placement) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement. The outcome is the change in arch length from baseline at each follow-up visit; larger absolute changes indicate greater relapse and worse post-treatment occlusal stability. Changes will be compared between the gold-plated and stainless-steel fixed-retainer groups.
Change in overjet | Baseline (T0, before retainer placement) and 1, 3, and 6 months (T1, T2, T3) after retainer placement.
  Overjet (mm) will be measured as the horizontal distance between the labial surface of the most prominent mandibular incisor and the palatal surface of the corresponding maxillary incisor, measured on study casts and/or intraoral records. Measurements will be taken at baseline (T0, before fixed-retainer placement) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement. The outcome is the change in overjet from baseline at each follow-up visit; larger absolute changes indicate greater relapse and worse post-treatment occlusal stability. Changes will be compared between the gold-plated and stainless-steel fixed-retainer groups.
Change in overbite | Baseline (T0, before retainer placement) and 1, 3, and 6 months (T1, T2, T3) after retainer placement.
  Overbite (mm) will be measured as the vertical overlap of the maxillary incisors over the mandibular incisors, using study casts and/or intraoral records. Measurements will be taken at baseline (T0, before fixed-retainer placement) and at 1 month (T1), 3 months (T2), and 6 months (T3) after retainer placement. The outcome is the change in overbite from baseline at each follow-up visit; larger absolute changes indicate greater relapse and worse post-treatment occlusal stability. Changes will be compared between the gold-plated and stainless-steel fixed-retainer groups.

CONTACTS AND LOCATIONS:
Overall Officials: NOOR NOOR, BDS, Principal Investigator — noor sattar
Locations (1):
- College of Dentistry, University of Baghdad - Orthodontic Clinics, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No